Analysis of hematoma morphology and related factors in patients with cerebral hemorrhage Prognosis Analysis of Different Treatment Schemes for Intracerebral Hemorrhage

Informed consent

Unit: Affiliated Hospital of Guizhou

Medical University

Submission date: March 9th, 2022

- 1. I agree to conduct clinical trials in strict accordance with the design and specific provisions of this protocol.
- 2. I understand that I can interrupt or terminate the clinical trial at any time in order to ensure the best interests of the subjects.
- 3. I agree that I will personally perform or supervise the clinical trial, and guarantee that all the researchers in my unit who assist me in performing the clinical trial are aware of their responsibilities in the clinical trial.
- 4. In the course of this clinical trial, I will strictly comply with the current QUM practices and the Declaration of Helsinki. And promised that the entire trial process will be consistent with ethical, ethical and scientific requirements
- 5. During the execution of clinical trials, I will strictly abide by all the laws and regulations related to clinical trials

Rights and interests of nursing subjects.

- 6. I promise that I will meet the EC requirements for review and approval.
- 7. I agree to maintain adequate and accurate medical records and to ensure that they are acceptable at any time

Inspections and inspections conducted by relevant laws and regulations.

8 I agree that any changes in clinical trial activities will be promptly reported to the Ethics Committee and involving subjects

Or other unexpected risk of unintended risk. In addition, I will not make any changes to the clinical trial protocol in clinical trial activities until the ethics committee approval, unless these modifications are made to reduce the risk of

| subjects in an emergency situation. | | |
|-------------------------------------|------------|-------|
| Name : | Signature: | Date: |